CLINICAL TRIAL: NCT01850329
Title: A Parental Educational Intervention to Facilitate Informed Consent for Pediatric Procedural Sedation in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Ko Lin (980425), Attending physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMUH-IRB- 980425
Record Dates: First submitted 2013-04-15; First posted 2013-05-09 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Informed Consent Process

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): No computed-assisted information program will be administered.
- intervention (Experimental): computed-assisted information program will be administered.
  Interventions: Other: computed-assisted information program

INTERVENTIONS:
Other: computed-assisted information program
  Arms: intervention

SUMMARY:
This study is planning to develop the computed-assisted information program and determine whether the computed-assisted information program are superior to routine discussion for informing parents in the emergency department (ED) about risks, benefits, and alternatives to receiving procedural sedation for their children.

ELIGIBILITY:
Inclusion Criteria:

* Parents with patients under 18 years of age
* patients receive the procedural sedation and anesthesia in the emergency department

Exclusion Criteria:

* clinically unstable
* refuse to participate
* unable to understand the consent process for this study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
structured questionnaire | before and immediately after the intervention when participants are in the emergency department, it is expected to take an expected average time of one hour
  a structured questionnaire with knowledge measure and satisfaction will be delivered to the participants for data collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung, Taiwan, Taiwan